CLINICAL TRIAL: NCT03038386
Title: Diagnostic Value of DECT Scan Compared to Diagnostic Needle Aspiration
Acronym: DEteCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meander Medical Center (Other)
Responsible Party: Principal Investigator, Mihaela Gamala, MD, Meander Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL54454.100.15
Record Dates: First submitted 2016-09-17; First posted 2017-01-31 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dual Energy CT (Other): In this study all patients undergo DECT scan to assess the value of DECT scan in diagnosing acute arthritis caused by gout. If the DECT scan demonstrates MSU depositions and the diagnosis of gout was not ascertained prior to DECT scanning by MSU crystals in the synovial fluid, then additional ultrasound guided aspiration will take place, with knowledge of DECT results, followed by repeat microscopy
  Interventions: Other: Dual Energy CT

INTERVENTIONS:
Other: Dual Energy CT — In this study all patients undergo DECT scan to assess the value of DECT scan in diagnosing acute arthritis caused by gout. If the DECT scan demonstrates MSU depositions and the diagnosis of gout was not ascertained prior to DECT scanning by MSU crystals in the synovial fluid, then additional ultrasound guided aspiration will take place, with knowledge of DECT results, followed by repeat microscopy

SUMMARY:
Rationale: Gout is a disease with growing incidence and complexity due to increased life expectancy, co-morbidity and medication. The disease can be diagnosed by microscopy, demonstrating monosodium uric acid (MSU) in synovial fluid of the affected joint or in tophi (subcutaneous or peritendinous MSU depositions). In daily practice, however, the diagnosis is difficult to ascertain due to sampling error (no synovial fluid acquired because the needle was not exactly placed in the affected joint, or the location of the gout might have been extra-articular e.g. around tendons) or to a different cause of acute arthritis (e.g. infection, reactive arthritis). Recently, Dual Energy CT scan has become available. This technique allows the visualization and quantification of MSU. Although imaging modalities such as DECT show promise in the classification of gout, the studies to date have been small and have primarily involved people with established disease.

A study with cross-sectional design in which patients for whom the clinical questions "does this patient have gout?" are referred for participation may contribute to assess the value of DECT scan in diagnosing acute arthritis caused by gout.

Objective: Assessment of value of DECT scan in diagnosing acute arthritis, caused by gout.

Study design: Prospective Study population: Patients with acute mono or oligo arthritis without prior diagnosis, the rheumatologist has an indication for diagnostic needle aspiration.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In current daily practice, patients with acute mono- or oligo-arthritis without prior diagnosis undergo a diagnostic aspiration of the affected joint. This can be done by blind aspiration or ultra sound guided aspiration depending on the judgement of the rheumatologist. The aspirated synovial fluid is then assessed by polarized microscopy to detect MSU crystals. The diagnostic value of DECT in acute gout attacks had not yet been established and is therefore not used in daily practice. In this study all patients undergo DECT scan to assess the value of DECT scan in diagnosing acute arthritis caused by gout. If the DECT scan demonstrates MSU depositions and the diagnosis of gout was not ascertained prior to DECT scanning by MSU crystals in the synovial fluid, then additional ultrasound guided aspiration will take place, with knowledge of DECT results, followed by repeat microscopy

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Mono or oligo arthritis (2-3 swollen joints)
* Indication for diagnostic aspiration of an inflamed joint in which gout is one of the possibilities

Exclusion Criteria:

* Polyarthritis ( up to 4 swollen joint);
* Chrystal proven gout in history
* Patient is on uric acid lowering therapy (Allopurinol, Benzbromaron, Febuxostat)
* Hip arthritis*
* Metal or prosthesis of the inflamed joint
* Highly suspicion of infectious arthritis
* Pregnancy
* Contra indication of joint aspiration (skin infection, hemophilia)
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity (95% CI) of DECT scanning for the detection of MSU deposits | 2 weeks

SECONDARY OUTCOMES:
clinical and laboratory predicators of positive DECT scan in patients with acute mono or oligo arthritis | 2 weeks
number of participants, in whom the first aspirate demonstrated no MSU and/or no synovial fluid, with MSU demonstrated after ultrasound guided joint aspiration | 2 weeks
number of participants with positive DECT lesions, in whom the first aspirate(s) demonstrated no MSU and/or no synovial fluid with MSU demonstrated after ultrasound guided joint aspiration at the place of positive DECT lesion | 2 weeks
cost of the gout diagnostic strategies (blind joint aspiration, ultrasound guided joint aspiration, DECT) will be calculated | 2 weeks
Patient satisfaction: What does the patient experience as the most patient-friendly way of diagnosing gout: DECT scan, ultrasound-guided joint aspiration or blind aspiration? | 2 weeks
  VAS DECT, blind joint aspiration, ultrasound guided joint aspiration
correlation between cardiovascular risk and the urate volume on DECT | 2 weeks
  correlation coefficient between cardiovascular risk (SCORE European and ACC/AHA) and the urate volume on DECT
number of patients with clinical diagnosis gout 6 and 12 month after het DECT | 6 and 12 month
number of patients on urate lowering medication 6 and 12 month after the DECT | 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Klaasen, MD, PhD, Principal Investigator — Meander Medical Center
Locations (1):
- Meander Medical Center, Amersfoort, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gamala M, Jacobs JWG, Linn-Rasker SF, Nix M, Heggelman BGF, Pasker-de Jong PCM, van Laar JM, Klaasen R. The performance of dual-energy CT in the classification criteria of gout: a prospective study in subjects with unclassified arthritis. Rheumatology (Oxford). 2020 Apr 1;59(4):845-851. doi: 10.1093/rheumatology/kez391. PMID 31504985